CLINICAL TRIAL: NCT06587282
Title: Multicenter, Single Arm Prospective, Non-Randomized Study Designed to Evaluate the Safety and Effectiveness of the BLOOM™ Micro-Occluder System for the Treatment of Patent Ductus Arteriosus (PDA) in Pre-mature Infants (PREEMIE)
Brief Title: PREEMIE: Study for Treatment of PDA in Premature Infants
Acronym: PREEMIE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Merit Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PDA-P3-23-01
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-08

CONDITIONS: Patent Ductus Arteriosus (PDA)
MeSH Terms: conditions — Ductus Arteriosus, Patent

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- PDA treatment (Experimental): PDA treated with Bloom Micro Occluder System
  Interventions: Device: Bloom Micro Occluder System

INTERVENTIONS:
Device: Bloom Micro Occluder System — Percutaneous transcatheter closure of PDA using Bloom Micro Occluder System

SUMMARY:
This multicenter, single arm, prospective, non-randomized study is designed to evaluate the safety and effectiveness of The Bloom Micro Occluder System for the treatment of patent ductus arteriosus (PDA) in pre-mature infants over a period of 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Subject is age ≥5 days at time of enrollment.
* Subject has a diagnosis of a hemodynamically significant patent ductus arteriosus (PDA) requiring closure.
* Subject has a PDA is ≤4.0 mm in diameter.
* Subject has a PDA is ≥5 mm in length.
* Subject's weight is between 600-2500 grams at time of enrollment.

Exclusion Criteria:

* Subject has pre-existing coarctation of the aorta.
* Subject has pre-existing left pulmonary artery stenosis.
* Subject has an Intracardiac thrombus that may interfere with the implant procedure
* Subject has other known hemodynamically significant congenital heart disease conditions at time of enrollment requiring intervention
* Subject has an active systemic infection at the time of enrollment.

Min Age: 5 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2025-03-06 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Safety Endpoint | 30 days
  Composite rate of device-related Major Adverse Events (MAE) of interest through 30 days following the index procedure.
Effectiveness Endpoint | 6 Months
  The rate of Clinical Success achieved at the 6-month follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Howaida El-Said, MD, Principal Investigator — Rady Children's Hospital
Locations (10):
- United States (10):
  - UC Davis Health, Sacramento, California
  - UC San Diego-Rady Children's Hospital, San Diego, California
  - Memorial Healthcare System-Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Washington University-St. Louis Children's Hospital, St Louis, Missouri
  - Nationwide Children's Hospital, Columbus, Ohio
  - Le Bonheur Children's Hospital, Memphis, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - Herma Heart Institute-Children's Wisconsin, Milwaukee, Wisconsin